CLINICAL TRIAL: NCT01876576
Title: The Impact of Diet Liberalization on Bowel Preparation for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 12D.247
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Colonic Diseases
Keywords: colonoscopy
MeSH Terms: conditions — Colonic Diseases | interventions — Lunch

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- clear liquids (Active Comparator): Clear liquids the day of bowel preparation up to 2.5 hrs before colonoscopy
  Interventions: Other: Clear liquids
- low residue diet (Active Comparator): Low residue breakfast and lunch up to 1pm; clear liquids thereafter up to 2.5 hrs before colonoscopy
  Interventions: Other: Low residue breakfast and lunch

INTERVENTIONS:
Other: Clear liquids — Clear liquids
  Arms: clear liquids
Other: Low residue breakfast and lunch — Low residue
  Arms: low residue diet

SUMMARY:
This study will evaluate the expansion of dietary options from clear liquids the entire day to a low reside breakfast and lunch for patients prior to undergoing bowel preparation with MoviPrep® and its effect on preparation quality for colonoscopy.

DETAILED DESCRIPTION:
This study will evaluate the expansion of dietary options from clear liquids the entire day to a low reside breakfast and lunch for patients prior to undergoing bowel preparation with MoviPrep® and its effect on preparation quality for colonoscopy. MoviPrep® is a commercially available 2 liter bowel purgative for use before colonoscopy in adults 18 years of age or older that is comprised of polyethylene glycol-electrolyte solution (PEG-ELS) plus sodium sulfate, sodium ascorbate, and ascorbic acid.

ELIGIBILITY:
Inclusion Criteria:

* Elective outpatients > 18 yrs undergoing colonoscopy

Exclusion Criteria:

* Unable or unwilling to give informed consent
* Age < 18 years
* Pregnant
* Breast feeding
* Gastroparesis - established or suspected
* Pseudo-obstruction - established or suspected
* Severe constipation (< 1 BM a week)
* Bowel obstruction
* Colon resection
* Chronic nausea or vomiting
* Known Glucose-6-Phosphate Dehydrogenase (G6PD) deficiency
* PEG allergy
* Significant psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Efficacy - Overall bowel cleansing based on Boston Bowel Preparation Scale score BBPS score of 2-3 for each segment AND total score | 1 day (At colonoscopy)

SECONDARY OUTCOMES:
Efficacy - Individual colon segment cleansing Successful cleansing defined as BBPS score of 2 - 3 for a segment | 1 day (At colonoscopy)

CONTACTS AND LOCATIONS:
Overall Officials: David Kastenberg, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States